CLINICAL TRIAL: NCT06530563
Title: the Efficacy and Safety of Oliceridine Fumarate Injection for Acute Pain After Abdominal Surgery: a Randomized, Double-blind, Positive-drug Parallel-controlled, Multi-center Clinical Study
Brief Title: the Efficacy and Safety of Oliceridine Fumarate Injection for Acute Pain After Abdominal Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Wu Jieping Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XiangyaHMZK
Record Dates: First submitted 2024-07-22; First posted 2024-07-31 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Acute Pain; Opioid Analgesic Adverse Reaction
Keywords: Oliceridine; acute pain after surgery; abdominal surgery
MeSH Terms: conditions — Acute Pain | interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oliceridine (Experimental): In the experimental group, the acute pain after surgery will be treated with Oliceridine, Dexmedetomidine, Ondansetron via patient controlled analgesia for 48 hours. Oliceridine 0.4-0.6mg/kg, Dexmedetomidine 2ug/kg, and Ondansetron 16mg will be supplied to 100ml analgesia pump, loading dose for 2ml, background infusion dose for 1-2ml/h, bolus for 2ml/ time, locked for 15min, maximum dose for 12ml/h.
  Interventions: Drug: Oliceridine Injection [Olinvyk]
- Sufentanil (Active Comparator): In the control group, the acute pain after surgery will be treated with Sufentanil, Dexmedetomidine, and Ondansetron via patient controlled analgesia for 48 hours. Sufentanil 2ug/kg , Dexmedetomidine 2ug/kg, and Ondansetron 16mg will be supplied to 100ml analgesia pump, loading dose for 2ml, background infusion dose for 1-2ml/h, bolus for 2ml/ time, locked for 15min, maximum dose for 12ml/h.
  Interventions: Drug: Sufentanil Citrate

INTERVENTIONS:
Drug: Oliceridine Injection [Olinvyk] — Oliceridine fumarate injection, specifications: 1mg/1mL, 2mg/2 mL, 10mg/10 mL; Stored in the dark, 15-30 ℃, not frozen; Jiangsu Nhwa pharmaceutical co., LTD. Production.
  Dexmedetomidine, specifications: 200ug/2ml; Ondansetron, specifications: 8mg/4ml.
  Other Names: Oliceridine fumarate injection; H20233508
  Arms: Oliceridine
Drug: Sufentanil Citrate — Sufentanil Citrate injection, specification: 50 ug/ml, 1 ml; Avoid light seal; Yichang humanwell pharmaceutical co., LTD.
  Dexmedetomidine, specifications: 200ug/2ml; Ondansetron, specifications: 8mg/4ml.
  Other Names: sufentanil injection
  Arms: Sufentanil

SUMMARY:
The goal of this clinical trial is to learn if Oliceridine fumarate injection works to treat acute pain after abdominal surgery. It will also learn about the safety of Oliceridine fumarate injection. The main questions it aims to answer are:

1. Does Oliceridine fumarate injection works to treat acute pain after abdominal surgery?
2. Does Oliceridine fumarate injection lead to less adverse effect?

Researchers will compare Oliceridine fumarate injection to a positive-drug (Sufentanil Citrate) to see if Oliceridine fumarate injection not inferior to sufentanil in the efficacy and safety for acute pain after abdominal surgery.

Participants will:

1. Receive patient controlled analgesia treat using Oliceridine or sufentanil after surgery
2. Be followed up every 6 hours until 48 hours after surgery or before discharge

DETAILED DESCRIPTION:
Traditional opioid, such as morphine, sufentanil , is an important drug treatment of postoperative period of acute pain, but their use is often limited because of significant side effects, such as respiratory depression, postoperative nausea and vomiting and sedation. If a drug is effective treatment of postoperative pain and avoid these adverse reactions, it will shorten the postoperative recovery time of patients, increase patients' satisfaction, and reduce hospitalization costs. Basic research shows that traditional opioids mainly bind to μ-opioid receptors and activate G protein signal transduction to exert analgesic effect. In addition, they stimulate the recruitment of β-arrestin, leading to respiratory depression, nausea and vomiting and other side effects. Oliceridine is a newly μ-opioid receptor agonist, which mainly activates the G protein signaling pathway to exert analgesic effect, but has a weak recruitment effect on β-arrestin and thus reduces the incidence of adverse reactions. However, due to its recent introduction to the market, there is still a lack of large-scale clinical studies on the application of Oliceridine in the population. So this topic to discuss the analgesic efficacy and adverse reactions of Oliceridine in patients with acute pain after abdominal surgery. Our study hypothesized that Oliceridine would have comparable analgesic efficacy and a lower incidence of associated side effects than sufentanil.

ELIGIBILITY:
Inclusion Criteria:

1.Preoperative inclusion criteria

1. aged ≥18 years and ≤75 years at screening;
2. Plan to undergo open or laparoscopic abdominal surgery, and the estimated operative time more than 2 hours.
3. able to understand and comply with research procedures and requirements, and can provide a written informed consent.

2.postoperative inclusion criteria:

1. patients who required open or laparoscopic surgery;
2. According to the investigator's judgment, the patient had recovered sufficiently from the intraoperative anesthesia protocol to accurately complete the protocol-specified questionnaire;

Exclusion Criteria:

1.preoperative exclusion criteria:

1. ASA grade >III
2. existing other acute or chronic pain conditions;
3. body mass index (BMI) < 18 or > 30 kg/m2;
4. with sleep apnea syndrome; 5 ) long-term opioid treatment, defined as receiving more than 15mg morphine equivalent units per day on more than 3 days per week for a period of more than 1 month in the 12 months prior to surgery;

6) suffering from mental or nervous system diseases (such as epilepsy, depression, schizophrenia, etc.), chronic obstructive pulmonary disease or pulmonary heart disease, heart failure, severe arrhythmia, etc; 7) with severe liver and kidney dysfunction; 8) Other conditions considered by the investigator to be inappropriate for enrollment.

Postoperative exclusion criteria:

1. intraoperative, postoperative or anesthetic deviations that may affect the efficacy and safety evaluation in the study;
2. evidence of hemodynamic instability or respiratory insufficiency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Area under the pain intensity time curve (AUC0-48, time in hours) in resting and moving states as assessed by numerical rating scale(NRS) during postoperative 48 hours | 48 hours
  Numerical rating scale(NRS), values from 0 to 10, 0 means "no pain", 10 means "the most intense pain", the higher score means a worse outcome; Area under the pain intensity time curve (AUC0-48), time in hours.

SECONDARY OUTCOMES:
Area under the pain intensity time curve (AUC) in resting and moving states as assessed by NRS during postoperative 12 hours and 24 hours. | 12 or 24 hours
  Area under the pain intensity time curve (AUC) in resting and moving states as assessed by NRS during postoperative 12 and 24 hours
total dose of rescue analgesics within 48 hours | 48 hours or the liquid of pump has run out before 48 hours.
  rescue analgesics include flurbiprofen axetil injection, parecoxib sodium and ketorolac tromethamine, reported in mg.
proportion of patients used rescue analgesics | 48 hours or when the liquid of pump has run out before 48 hours.
  proportion of patients used rescue analgesics
Incidence of respiratory depression | 48 hours
  Incidence of respiratory depression (i.e., respiratory rate ≤8 breaths/minute or oxygen saturation (SpO2)<90%)
The occurrence of nausea and vomiting | 48 hours
  The proportion of patients with nausea and vomiting within 48 hours and the proportion of patients using antiemetic drugs. Antiemetic drugs (i.e., ondansetron or tropisetron) report in mg.
Condition of sedation | 48 hours
  Condition of sedation is assessed by observer's assessment alert/Sedation(OAA/S), value from 0 to 5, grade 0 means deep sedation, grade 5 means fully awake.
the occurrence of adverse events | 1 month
  the occurrence of adverse events
Satisfaction scores within 48 h of the participants and researchers | 48 hours
  Satisfaction scores grade from 1 to 5. 5 means very satisfied, 4 means satisfied, 3 means general satisfied, 2 means not satisfied, 1 means very dissatisfied.
the use of Antiemetic drugs | 48 hours
  the use of antiemetic drugs.
the score of quality of recovery-15 items | 48 hours
  the score of quality of recovery-15 items(QoR-15)

OTHER OUTCOMES:
the analgesic effect and adverse reactions of Oliceridine in preoperative and postoperative hypertensive patients taking angiotensin-converting enzyme inhibitor/angiotensin receptor blocker(ACEI/ARB) drugs | 1 month
  the analgesic effect include the area under the pain intensity time curve (AUC, time in hours) in resting and moving states as assessed by numerical rating scale(NRS) at 12, 24 and 48 hours, the proportion of using rescue analgesics. The adverse reactions include the proportion of patients with nausea and vomiting within 48 hours and the proportion of patients using antiemetic drugs, the incidence of respiratory depression and the condition of sedation assessed by observer's assessment alert/Sedation(OAA/S).

CONTACTS AND LOCATIONS:
Overall Officials: e wang, doctor, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No